CLINICAL TRIAL: NCT02971696
Title: Sorafenib Versus Best Supportive Care in Egyptian Hepatocellular Carcinoma Patients. Prospective Phase III Study
Brief Title: Sorafenib Versus Best Supportive Care in Egyptian Hepatocellular Carcinoma Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Noha El Baghdady, Ph.D Candidate, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 40
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: HCC
MeSH Terms: interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HCC patients (Group 1) (Experimental): Sorafenib will be administrated at a dose of 400 mg twice daily (consisting of two 200-mg tablets).Treatment interruptions and up to two dose reductions (first to 400 mg once daily and then to 400 mg every 2 days) will permitted for drug- related adverse effects. If further dose reductions will required, patients will withdraw from the study
  Interventions: Drug: Sorafenib
- HCC patients (Group 2) (Active Comparator): Patient will take best supportive care
  Interventions: Drug: Best Supportive care

INTERVENTIONS:
Drug: Sorafenib — Sorafenib will be administrated at a dose of 400 mg twice daily (consisting of two 200-mg tablets).Treatment interruptions and up to two dose reductions (first to 400 mg once daily and then to 400 mg every 2 days) will permitted for drug- related adverse effects. If further dose reductions will required, patients will withdraw from the study
  Other Names: nexavar
  Arms: HCC patients (Group 1)
Drug: Best Supportive care — Liver Support, pain management
  Other Names: Liver Support
  Arms: HCC patients (Group 2)

SUMMARY:
The aim of the study is to evaluate the efficacy of sorafenib, compared to the best supportive care (BSC), in two cohorts of patients who presented with advanced hepatocellular carcinoma (HCC) based on etiology of hepatitis C virus.

DETAILED DESCRIPTION:
In Egypt, chronic hepatitis C virus (HCV) infection occurs in around 10% of the population (about 8 million individuals), and is a leading cause of liver cirrhosis, hepatocellular carcinoma, and mortality. Although HCV genotype 4 constitutes about 20% of HCV infections worldwide, the prevalence in Egypt is more than 90%.(Waked et al., 2016)

In 2014 Omar et al. reviewed 41 patients in a study to evaluate Sorafenib for Egyptian patients with advanced hepatocellular carcinoma at a median follow up period of 13 months, the median PFS for the whole group was 4 months; the median OS for the whole group is 6.25 months.(Abdel-Rahman et al., 2014)

Till current, no studies have evaluated the Sorafenib efficacy in comparison to the best supportive care treatment in HCC patients whose etiology from HCV genotype 4 ( the most prevalent hepatitis C virus genotype in Egypt).

So, The study aims to evaluate the efficacy of sorafenib, compared to the best supportive care (BSC), in two cohorts of patients who presented with advanced hepatocellular carcinoma (HCC) based on etiology of hepatitis C virus.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age
2. Patients based on etiology of hepatitis C virus.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or less
4. Child-Pugh liver function class A,B
5. A life expectancy of 12 weeks or more
6. adequate hematologic function (platelet count, ≥60×109 per liter; hemoglobin, ≥8.5 g per deciliter; and prothrombin time international normalized ratio, ≤2.3; or prothrombin time, ≤6 seconds above control), adequate hepatic function (albumin, ≥2.8 g per deciliter; total bilirubin, ≤3 mg per deciliter [51.3 µmol per liter]; and alanine aminotransferase and aspartate aminotransferase, ≤5 times the upper limit of the normal range), and adequate renal function (serum creatinine, ≤1.5 times the upper limit of the normal range).
7. Patients were required to have at least one untreated target lesion that could be measured in one dimension, according to the Response Evaluation Criteria in Solid Tumors (RECIST)

Exclusion Criteria:

1. Had previously received molecularly targeted therapies or any other systemic treatment.
2. Any co morbid disease that will confuse the assessment of the Quality of life questionnaire scoreFHSI-8 score.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | 12 months
  Overall survival is defined as the duration from the start of treatment date till date of last contact or death date.
Event free survival | 12 months
  Event free survival was defined as the duration from the date of diagnosis till the date of first event (death, radiological progression, symptomatic progression) or the date of last contact if the patient did not develop the event.

SECONDARY OUTCOMES:
Detection of changes in quality of life | 12 months
  through application of QLQ FHSI-8 questionnaire every two months in both arms
Sorafenib induced side effects | 12 months
  incidence and severity

CONTACTS AND LOCATIONS:
Overall Officials: AbdelRahman Elnaggar, Prof., Study Chair — MTI University
Locations (3):
- Egypt (3):
  - El Kahraba Hosital, Cairo, N/A = Not Applicable
  - Ain Shams University Hospital, Cairo
  - Nasser Institute, Cairo

IPD SHARING:
Plan to Share IPD: No